CLINICAL TRIAL: NCT06929182
Title: OBServaToIre National Des Patients AnTiphospholipidEs traités Par Anticoagulants Oraux Directs
Brief Title: OBServaToIre interNational Des Patients AnTiphospholipidEs traités Par Anticoagulants Oraux Directs
Acronym: OBSTINATE 2
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Virginie Dufrost, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2025PI048
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Antiphospholipid Syndrome (APS); Direct Oral Anticoagulants (DOACs); Thrombotic and Bleeding Events; Safety
Keywords: safety of DOACs; "non-high risk" APS patients; Observatory; Phase IV; International
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Population of "non-high risk" thrombotic APS patients treated with DOAC: Non-high-risk" APS is defined by the absence of a history of arterial or microcirculatory thrombosis, the absence of valvulopathy related to APS, and a biological profile with only one or two positive antiphospholipid tests
  Interventions: Other: "non-high risk" thrombotic APS patients treated with DOAC

INTERVENTIONS:
Other: "non-high risk" thrombotic APS patients treated with DOAC — There is no specific intervention in this study. Routine care data will be collected from patients with a 'non-high-risk' APS profile who are currently being treated with DOACs or have been in the past.

SUMMARY:
This registry will make it possible to collect large-scale data on SAPL patients, particularly those treated with DOACs, in order to better assess the frequency of thrombotic and hemorrhagic events in this population of "non-high-risk" thrombotic SAPL patients treated with DOACs. The results will help refine treatment recommendations and could form the basis of future clinical trials.

In this study, there will be no modification of the usual care and no additional follow-up. Follow-up will be carried out during the patient's usual visits in the context of his or her pathology, the frequency of which will be left to the discretion of the usual physician. No additional consultations/hospitalizations/examinations will be carried out as part of the study. Data normally recorded in the medical record will be collected over a 5-year period, in line with standard patient follow-up.

DETAILED DESCRIPTION:
Direct oral anticoagulants (DOACs) are indicated as first-line therapy for the prevention of recurrence of venous thromboembolism. The management of APS patients is based on long-term anticoagulation, which the gold standard vitamin K antagonist (VKA) including warfarin. Managing VKA is sometimes a challenge in these patients due to their young age and prolonged treatment requiring regular monitoring of INR and numerous drug interactions. DOACs don't require biological monitoring so would represent a potential easier oral treatment for these APS patients.

In 2016, the first controlled randomized compared DOACs vs VKA in about fifty APS patients (RAPS study) using biological data (generation of thrombin). The safety profile (thrombotic recurrence / hemorrhage) seemed reassuring; However, the duration of follow-up and the number of included subjects were insufficient to conclude on clinical safety criteria.

Subsequently, case series have reported the use of DOACs in these patients. Thus, a meta-analysis on individual data covering all of the literature and including these case series was recently published: 447 APS patients treated with DOACs were included and for the first time, a rate of 16% recurrent thrombosis has been identified despite treatment. This recurrence rate is abnormally high compared to that with VKA. Some risk factors for recurrent thrombosis have been identified: the positivity of all antiphospholipid biological tests ("triple positivity"; OR = 4.3 [95% CI; 2.3-7.7]), and in patients treated with anti-Xa only (rivaroxaban or apixaban), a history of arterial thrombosis was associated with a higher risk of thrombotic recurrence (32% vs 14%, p = 0.006).

These results were confirmed by the TRAPS trial, which had to be prematurely stopped due to an excess of thrombotic events in the group of 59 "triple positive" APS patients treated with rivaroxaban (12% vs 0%) compared to the group treated with warfarin.

Thus, the use of DOACs does not appear to be risk free in all patients with APS, particularly those with "triple positivity" or those with a history of arterial thrombosis who represent a group of patients at "high risk" thrombosis.

The European Medicines Agency (EMA) has diffused a letter recommending against the use of DOACs in patients with APS, especially triple-positive patients, and the use of VKAs has to be considered. It is important to emphasize that this modification does not constitute a contraindication to the use of DOACs but a recommendation.

For the other "non-high risk" APS patients who constitute the majority of APS patients, we have not strong arguments to justify a routine DOACs-VKA switch. Commonly in these patients, DOACs treatment was started in the acute phase of a thrombotic episode, before the diagnosis of APS was made. According to international recommendations, to conclude for an APS, it is necessary to control the aPL laboratory tests twice at least 3 months apart to conclude that there is persistent positivity. Thus the diagnosis of APS is often made several months after the thrombotic event and therefore several months after the introduction of anticoagulant treatment.

Taking into account the advantages on the quality of life of DOACs compared to VKAs, patients are often not in favor of modifying their anticoagulant treatment, especially if it has been started for many years with good tolerance. In addition, the switch from one well-balanced anticoagulant treatment to another is not without risk in terms of thrombosis or bleeding. It is for these reasons that a number of patients with APS remain on DOACs.

On the other hand, the European League Against Rheumatism (EULAR) recommends - in its recommendations for the APS management published on May 15, 2019 - to contraindicate the use of rivaroxaban in "high risk" APS patients but does not position itself in relation to the use of other DOACs or in "non-high risk" patients. In these patients, treatment could be continued and their follow-up would then become crucial to confirm that "non-high risk" patients are indeed at low risk of recurrent thrombosis.

For these "non-high risk" patients currently treated with DOACs, we do not currently have follow-up data on a sufficient group of patients. Therefore, it becomes urgent to collect in an exhaustive and prospective manner, all the data of "non-high risk" APS patients treated with DOACs and until then not monitored. The results will make it possible to better identify the target population that could benefit from this type of treatment. The results would also help prevent unnecessary VKA relays that carry their own risks.

ELIGIBILITY:
Inclusion Criteria:

* Person having received complete information on the organization of the research and not having opposed the use of this data
* Male or female aged 18 and over;
* Carrier of a thrombotic APS according to the Sydney classification criteria, regardless of the length of time in the disease
* Having received a direct oral anticoagulant (DOAC) treatment which is currently discontinued.
* Or currently treated with DOAC

Exclusion Criteria:

* Incomplete Sydney classification criteria
* Presence of a triple antiphospholipid positivity
* History of arterial thrombosis
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the French Public Health Code:

  * Pregnant, parturient or nursing mother
  * Minor person (not emancipated)
  * Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
  * Person of full age unable to express consent
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric treatment under Articles L. 3212-1 and L. 3213-1 of the French Public Health Code.
* Signature of the research participation opposition form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of "non-high-risk" thrombotic SAPL patients treated with DOACs. Given current recommendations, SAPL patients at "high risk" of thrombosis (triple positivity, history of arterial thrombosis) should not be treated with DOACs and will not be included.
  Recruitment will be carried out via the departments authorized to manage these patients, at the time of their consultation or hospitalization. Patients will be invited to participate in the study as part of their regular follow-up visit.
  Services: services authorized to care for these patients within the open international investigator hospitals
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2035-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of thrombotic complications | From enrollment to the thrombotic recurrence or the end of the study (5 years post-inclusion)
  Occurrence of thrombotic recurrence within 5 years of inclusion confirmed by a reference examination :
  * PE: CT angiography, ventilation / perfusion scintigraphy
  * Stroke: MRI or brain scan
  * Venous or peripheral arterial thrombosis: Doppler ultrasound, CT angiography, MRI
  * MI or cardiac microcirculatory impairment: ECG and troponin, coronary angiography, TTE, MRI
  * Skin: skin biopsy
  * Adrenal or intra-alveolar hemorrhage: CT scan or MRI

SECONDARY OUTCOMES:
Risk Factors of thrombotic recurrence | From enrollment to the thrombotic recurrence or the end of the study (5 years post-inclusion)
  Occurrence of a venous, arterial or microcirculatory thrombotic recurrence confirmed by a baseline examination (detailed in the primary endpoint)
Frequency of manifestations associated with APS (non-criteria manifestations according to the Sydney classification criteria) | From enrollment to the thrombotic recurrence or the end of the study (5 years post-inclusion)
  Occurrence of non-criteria manifestations according to the Sydney criteria: thrombocytopenia, hemolytic anemia, valve disease, livedo, nephropathy due to APS, superficial venous thrombosis, chorea
Frequency of hemorrhages and other adverse events | From enrollment to the thrombotic recurrence or the end of the study (5 years post-inclusion)
  Occurrence of hemorrhagic accident according to the definition of the International Society on Thrombosis and Haemostasis

CONTACTS AND LOCATIONS:
Overall Officials: Virginie DUFROST, MD, Principal Investigator — CHRU - Nancy
Locations (1):
- Vall d´Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pengo V, Denas G, Zoppellaro G, Jose SP, Hoxha A, Ruffatti A, Andreoli L, Tincani A, Cenci C, Prisco D, Fierro T, Gresele P, Cafolla A, De Micheli V, Ghirarduzzi A, Tosetto A, Falanga A, Martinelli I, Testa S, Barcellona D, Gerosa M, Banzato A. Rivaroxaban vs warfarin in high-risk patients with antiphospholipid syndrome. Blood. 2018 Sep 27;132(13):1365-1371. doi: 10.1182/blood-2018-04-848333. Epub 2018 Jul 12. PMID 30002145
- [Background] Dufrost V, Risse J, Reshetnyak T, Satybaldyeva M, Du Y, Yan XX, Salta S, Gerotziafas G, Jing ZC, Elalamy I, Wahl D, Zuily S. Increased risk of thrombosis in antiphospholipid syndrome patients treated with direct oral anticoagulants. Results from an international patient-level data meta-analysis. Autoimmun Rev. 2018 Oct;17(10):1011-1021. doi: 10.1016/j.autrev.2018.04.009. Epub 2018 Aug 11. PMID 30103045
- [Background] Cohen H, Hunt BJ, Efthymiou M, Arachchillage DR, Mackie IJ, Clawson S, Sylvestre Y, Machin SJ, Bertolaccini ML, Ruiz-Castellano M, Muirhead N, Dore CJ, Khamashta M, Isenberg DA; RAPS trial investigators. Rivaroxaban versus warfarin to treat patients with thrombotic antiphospholipid syndrome, with or without systemic lupus erythematosus (RAPS): a randomised, controlled, open-label, phase 2/3, non-inferiority trial. Lancet Haematol. 2016 Sep;3(9):e426-36. doi: 10.1016/S2352-3026(16)30079-5. PMID 27570089